CLINICAL TRIAL: NCT05515835
Title: Relationship Between Effect Duration of Rocuronium and Body Composition Analysis Data.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Prof., Samsung Medical Center
Other Study IDs: SMC 2022-07-160
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Rocuronium; Body Composition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rocuronium: The patient will be given 50mg of rocuronium intravenously for induction.
  Interventions: Device: body composition analysis

INTERVENTIONS:
Device: body composition analysis — Patients will undergo body composition analysis using bioelectical impedance method before anesthesia.

SUMMARY:
The induction dose of rocuronium is typically decided based on the patient's body weight, but the effect duration of rocuronium is variable. Some studies suggest that body composition analysis data, such as skeletal muscle mass or total body water, may correlate better with the duration time of rocuronium. Therefore, we plan to analyse body composition in patients undergoing total intravenous general anesthesia, give the patients a fixed dose (50mg) of rocuronium, and check the correlation between duration time of rocuronium and body composition analysis data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ASA class I-II undergoing total intravenous general anesthesia

Exclusion Criteria:

* too overweight (over 111.11kg, which corresponds to less than 0.45mg/kg of induction dose of rocuronium)
* too underweight (under 41.67kg, which corresponds to more than 1.2mg/kg of induction dose of rocuronium)
* pregnancy
* prediagnosed muscle or nerve related disease
* unsuitable for body composition analysis using bioelectrical impedance method
* unsuitable for neuromuscular block monitoring

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ASA class I-II undergoing total intravenous general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
time to TOF1 | up to 1 hour after rocuronium administration during induction of anesthesia
  correlation between the time from induction to recovery of 1st TOF twitch and age, sex, ASA class, body weight, and body composition analysis data
time to TOF4 | up to 1.5 hour after rocuronium administration during induction of anesthesia
  correlation between the time from induction to recovery of 4th TOF twitch and age, sex, ASA class, body weight, and body composition analysis data

SECONDARY OUTCOMES:
time to loss of TOF | up to 5 minutes after rocuronium administration during induction of anesthesia
  correlation between the time from injection of rocuronium to complete loss of TOF twitch and age, sex, ASA class, body weight, and body composition analysis data

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University, School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided